CLINICAL TRIAL: NCT03880032
Title: Happy Mother-Healthy Baby: An Anxiety-focused Early Prenatal Intervention for the Prevention of Common Mental Disorders in Pakistan
Brief Title: Happy Mother-Healthy Baby: An Anxiety-focused Early Prenatal Intervention
Acronym: HMHB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Human Development Research Foundation, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH111859-01 (NIH)
Record Dates: First submitted 2019-03-04; First posted 2019-03-19 (Actual); Results first posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Postpartum Depression; Small for Gestational Age at Delivery; Preterm Birth; Anxiety; Birth Weight
Keywords: anxiety; depression; birth outcomes
MeSH Terms: conditions — Depression, Postpartum; Premature Birth; Anxiety Disorders; Birth Weight; Depression

STUDY DESIGN:
Intervention Model Description: Women with at least mild anxiety but not depression will be enrolled simultaneously into an intervention or an enhanced usual care group during pregnancy. Women in the intervention group will receive individual-based cognitive behavioral therapy. Women in the control group with receive enhanced usual care.
Who Masked: Investigator, Outcomes Assessor
Masking Description: To maintain masking during the trial, intervention and assessment teams will not have any interaction during the trial, as they will be placed at separate locations within the Obstetrics Department of Holy Family Hospital (HFH). Furthermore, participants will be instructed not to disclose which type of treatment they are receiving to the assessment team. Fidelity of masking will be measured by having assessors guess the trial arm of each participant at the end of follow-up assessment. We hypothesize that assessors will only be able to correctly guess the condition of participants at a chance rate of nearly 50% at follow-up assessments, indicating that masking is maintained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy Intervention for Anxiety (Experimental): Pregnant women experiencing anxiety randomized to the Happy Mother Healthy Baby (HMHB) intervention receive a CBT-based psychosocial intervention (with six core and up to six booster sessions). HMHB is a facility-based intervention delivered by non-specialist providers. It is aimed to raise psychosocial awareness and facilitate positive change inter personal wellbeing, social support, and bonding with their baby during pregnancy. It addresses with relapse prevention, planning for the baby's arrival, and in management of emotional challenges in the early postnatal period. Family member/s will be invited to attend 3 core sessions.
  Interventions: Behavioral: Cognitive Behavioral Therapy Intervention for Anxiety
- Enhanced Usual Care (No Intervention): Women randomized to the control group will receive enhanced usual care (EUC). The World Health Organization (WHO) recommends 8 antenatal visits for a positive pregnancy experience, the number of visits our EUC control group participants will receive (depending on their gestational week). Usual care will also be enhanced by hospital staff receiving additional training in mental health treatment and counseling. Reminder calls were given, provider visits were facilitated (shorter wait times), and transportation to assist participants in attending appointments and medically indicated ultrasounds were paid for (as in the intervention group).

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy Intervention for Anxiety — Happy Mother Healthy Baby (HMHB) is a CBT-based psychosocial intervention for expectant women experiencing anxiety during their pregnancy. Strategies such as empathetic listening, thought challenging, behavior activation, problem management, take-home exercises, and family involvement are employed by HMHB.
  Arms: Cognitive Behavioral Therapy Intervention for Anxiety

SUMMARY:
In the proposed study the investigators will develop an early prenatal preventive intervention targeting anxiety and conduct a randomized controlled trial in Pakistan to test its efficacy in reducing generalized anxiety disorder and major depression in mothers in late pregnancy and the postnatal period. Investigators will evaluate the impact of the intervention on fetal and infant growth restriction as well as examine how the impact of the intervention is mediated (to elucidate mechanisms) and/or modified (to help optimize future adaptations of the program) by various social factors. A cost-effectiveness evaluation will shed light on the costs and benefits of intervention components in relation to outcomes, enabling policy-makers and public health planners to scale up this intervention according to resource budgeting requirements.

DETAILED DESCRIPTION:
Common mental disorders (CMDs) such as anxiety and depression occur frequently in pregnancy and the postnatal period in lower- and middle income countries (LMICs). Prenatal anxiety, both subthreshold and clinical, adversely affects maternal wellbeing and outcomes among offspring, and is a major predictor of subsequent depression. Preventive approaches have enormous potential to reduce the negative effects of postnatal mental disorders in mothers and improve child outcomes. The study team proposes to create a scalable and sustainable early prevention intervention focusing on anxiety symptoms in pregnant women, to be delivered by non-specialist providers (Aim 1). The investigators will evaluate this preventive intervention through a trial by randomizing 1200 pregnant women from a public hospital in Islamabad Pakistan to either our Cognitive Behavioral Therapy-based (CBT-based) early-in-pregnancy program or to usual care. The investigators will study the effects of the intervention on 1) CMDs in the 3rd trimester of pregnancy and at 6 weeks postpartum (Aim 2) and on 2) fetal and newborn small-for-gestational age (SGA) outcomes (Aim 3). The investigators will also examine if interpersonal violence, perceived stress and social support mediate and/or modify the intervention effects on CMDs and perinatal outcomes (Aim 4). Finally, the investigators will conduct a cost-effectiveness evaluation, comparing costs and healthcare utilization for women in the prenatal intervention and enhanced usual care groups (Aim 5). Focusing on anxiety reduction is a major innovation; anxiety has not been addressed within prenatal intervention packages in LMICs, despite its association with increased postpartum depression and suboptimal fetal and infant outcomes. Pakistan has high prevalence of both women with prenatal anxiety (35% to 49%) and SGA newborns (~47%), providing an ideal research opportunity. The CBT-based approach, appropriate given its indication for anxiety and depression, is grounded in preliminary work in this population, where the investigators have previously successfully reduced postpartum depression. Intervening early in pregnancy is a further innovation that is critical for building the evidence base for preventative approaches to reduce maternal CMDs and related perinatal outcomes. The proposed mediation and effect modification analyses will improve understanding of mechanism(s) of action and help identify subpopulations for programmatic targeting. The use of non-specialized providers and integration within the primary care environment will guide scale up, while incorporating a cost-effectiveness analysis will aid policy-makers in resource allocation decisions. This study will inform the integration of preventive strategies that target anxiety with existing approaches for treatment of perinatal depression to further the evidence-base for transdiagnostic mental health initiatives globally, and will inform policies to support lifelong maternal mental health and resilience across generations

ELIGIBILITY:
Inclusion Criteria:

1. ability to understand spoken Urdu
2. pregnant, ≤22 weeks' gestation
3. age ≥18 years
4. residence ≤20 km of Holy Family Hospital
5. intent to reside in the study areas until the completion of the study
6. score ≥8 for anxiety on the Hospital Anxiety and Depression Scale (HADS)

Exclusion Criteria:

1. Current major a depressive episode (MDE on SCID) or life-threatening health conditions including e.g. active severe depression or suicidal ideation
2. Self-report of past or current significant learning disability
3. Self-report of past or current psychiatric disorder (e.g. bipolar disorder or schizophrenia) or psychiatric care (e.g. current use of anxiolytic drug and/or other psychotropic drug)
4. medical disorders or severe maternal morbidity that require inpatient management that would preclude participation (101)
5. ICU admission indicated by diagnosis (not only for assessment)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela J. Surkan, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Holy Family Hospital, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified project data from the study will be posted on ClinicalTrials.gov and the National Institute of Mental Health (NIMH) data archive.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol and statistical analysis plan (SAP) have been shared in the study protocol paper published in BMJ Open (PMID: 32300002; PMCID: PMC7200036). The Informed Consent Forms (ICF) have been published accessed and as the Supplementary Material associated with that article.
Access Criteria: There is a link to the Informed Consent Forms (ICF) on the open access website for our protocol paper. Please see: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7200036/

REFERENCES:
- [Background] Surkan PJ, Hamdani SU, Huma ZE, Nazir H, Atif N, Rowther AA, Chaudhri R, Zafar S, Mullany LC, Malik A, Rahman A. Cognitive-behavioral therapy-based intervention to treat symptoms of anxiety in pregnancy in a prenatal clinic using non-specialist providers in Pakistan: design of a randomised trial. BMJ Open. 2020 Apr 15;10(4):e037590. doi: 10.1136/bmjopen-2020-037590. PMID 32300002
- [Background] Rowther AA, Kazi AK, Nazir H, Atiq M, Atif N, Rauf N, Malik A, Surkan PJ. "A Woman Is a Puppet." Women's Disempowerment and Prenatal Anxiety in Pakistan: A Qualitative Study of Sources, Mitigators, and Coping Strategies for Anxiety in Pregnancy. Int J Environ Res Public Health. 2020 Jul 8;17(14):4926. doi: 10.3390/ijerph17144926. PMID 32650551
- [Background] Rauf N, Zulfiqar S, Mumtaz S, Maryam H, Shoukat R, Malik A, Rowther AA, Rahman A, Surkan PJ, Atif N. The Impact of the COVID-19 Pandemic on Pregnant Women with Perinatal Anxiety Symptoms in Pakistan: A Qualitative Study. Int J Environ Res Public Health. 2021 Aug 4;18(16):8237. doi: 10.3390/ijerph18168237. PMID 34443987
- [Background] Kazi AK, Rowther AA, Atif N, Nazir H, Atiq M, Zulfiqar S, Malik A, Surkan PJ. Intersections between patient-provider communication and antenatal anxiety in a public healthcare setting in Pakistan. PLoS One. 2021 Feb 5;16(2):e0244671. doi: 10.1371/journal.pone.0244671. eCollection 2021. PMID 33544747
- [Background] Nazir H, Rowther AA, Rauf N, Atiq M, Kazi AK, Malik A, Atif N, Surkan PJ. 'Those whom I have to talk to, I can't talk to': Perceived social isolation in the context of anxiety symptoms among pregnant women in Pakistan. Health Soc Care Community. 2022 Nov;30(6):e5885-e5896. doi: 10.1111/hsc.14019. Epub 2022 Sep 19. PMID 36121172
- [Background] Zaidi A, Khan A, Rowther A, Nazir H, Perin J, Rauf N, Mumtaz S, Naseem H, Atif N, Rahman A, Surkan PJ, Malik A. Cultural adaptation and psychometric validation of the Pregnancy Experience Scale-Brief version (PES-Brief) in Pakistani women with antenatal anxiety symptoms. SSM Ment Health. 2022 Dec;2:100055. doi: 10.1016/j.ssmmh.2021.100055. Epub 2021 Dec 24. PMID 36969715
- [Background] Atif N, Rauf N, Nazir H, Maryam H, Mumtaz S, Zulfiqar S, Shouket R, Rowther AA, Malik A, Rahman A, Surkan PJ. Non-specialist-delivered psychosocial intervention for prenatal anxiety in a tertiary care setting in Pakistan: a qualitative process evaluation. BMJ Open. 2023 Feb 23;13(2):e069988. doi: 10.1136/bmjopen-2022-069988. PMID 36822801
- [Background] Malik A, Park S, Mumtaz S, Rowther A, Zulfiqar S, Perin J, Zaidi A, Atif N, Rahman A, Surkan PJ. Perceived Social Support and Women's Empowerment and Their Associations with Pregnancy Experiences in Anxious Women: A Study from Urban Pakistan. Matern Child Health J. 2023 May;27(5):916-925. doi: 10.1007/s10995-023-03588-6. Epub 2023 Feb 6. PMID 36746839
- [Result] Atif N, Nazir H, Zafar S, Chaudhri R, Atiq M, Mullany LC, Rowther AA, Malik A, Surkan PJ, Rahman A. Development of a Psychological Intervention to Address Anxiety During Pregnancy in a Low-Income Country. Front Psychiatry. 2020 Jan 10;10:927. doi: 10.3389/fpsyt.2019.00927. eCollection 2019. PMID 31998151
- [Derived] Siebach KF, Park S, Mansoor M, Atif N, Zaidi A, Rahman A, Malik A, Surkan PJ. The Association of Spousal Relationship Quality and Social Support With Maternal-Infant Bonding: Moderating Roles of Maternal Age and Paternal Occupation. Infancy. 2025 Jan-Feb;30(1):e12647. doi: 10.1111/infa.12647. PMID 39740193
- [Derived] Surkan PJ, Park S, Sheng Z, Zaidi A, Atif N, Osborne LM, Rahman A, Malik A. Effects of a Prenatal Anxiety Randomized Controlled Trial Intervention on Infant Development in Pakistan. Acad Pediatr. 2025 Jan-Feb;25(1):102551. doi: 10.1016/j.acap.2024.07.018. Epub 2024 Aug 2. PMID 39097000
- [Derived] Nisar A, Xiang H, Perin J, Malik A, Zaidi A, Atif N, Rahman A, Surkan PJ. Impact of an intervention for perinatal anxiety on breastfeeding: findings from the Happy Mother-Healthy Baby randomized controlled trial in Pakistan. Int Breastfeed J. 2024 Aug 2;19(1):53. doi: 10.1186/s13006-024-00655-8. PMID 39095863
- [Derived] Siebach KF, Perin J, Malik A, Atif N, Zaidi A, Rahman A, Surkan PJ. Results of a cognitive behavior therapy-based intervention for antenatal anxiety on birth outcomes in Pakistan: a randomized control trial. Sci Rep. 2024 Jun 14;14(1):13806. doi: 10.1038/s41598-024-64119-z. PMID 38877077
- [Derived] Sun Y, Park S, Malik A, Atif N, Zaidi A, Rahman A, Surkan PJ. Pregnancy stressors and postpartum symptoms of depression and anxiety: the moderating role of a cognitive-behavioural therapy (CBT) intervention. Gen Psychiatr. 2024 Feb 28;37(1):e101136. doi: 10.1136/gpsych-2023-101136. eCollection 2024. PMID 38440406
- [Derived] Surkan PJ, Malik A, Perin J, Atif N, Rowther A, Zaidi A, Rahman A. Anxiety-focused cognitive behavioral therapy delivered by non-specialists to prevent postnatal depression: a randomized, phase 3 trial. Nat Med. 2024 Mar;30(3):675-682. doi: 10.1038/s41591-024-02809-x. Epub 2024 Feb 16. PMID 38365951
- [Derived] Sherer ML, Malik A, Osborne LM, Rowther AA, Zaidi A, Atif N, Rahman A, Kahloon LE, Salman M, Yenokyan G, Surkan PJ. Biological Mechanisms in Pregnant Women With Anxiety (Happy Mother-Healthy Baby Supplement Study): Protocol for a Longitudinal Mixed Methods Observational Study. JMIR Res Protoc. 2023 Apr 11;12:e43193. doi: 10.2196/43193. PMID 37040167
- [Derived] Yonemoto N, Nagai S, Mori R. Schedules for home visits in the early postpartum period. Cochrane Database Syst Rev. 2021 Jul 21;7(7):CD009326. doi: 10.1002/14651858.CD009326.pub4. PMID 34286512

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Behavioral Therapy (CBT) Intervention for Anxiety: Pregnant women experiencing anxiety randomized to the Happy Mother Healthy Baby (HMHB) intervention receive a CBT-based psychosocial intervention (with six core and up to six booster sessions). HMHB is a facility-based intervention delivered by non-specialist providers. It is aimed to raise psychosocial awareness and facilitate positive change inter personal wellbeing, social support, and bonding with their baby during pregnancy. It addresses with relapse prevention, planning for the baby's arrival, and in management of emotional challenges in the early postnatal period. Family member/s will be invited to attend 3 core sessions.
  Cognitive Behavioral Therapy Intervention for Anxiety: Happy Mother Healthy Baby (HMHB) is a CBT-based psychosocial intervention for expectant women experiencing anxiety during their pregnancy. Strategies such as empathetic listening, thought challenging, behavior activation, problem management, take-home exercises, and family involvement are employed by HMHB.
- Enhanced Usual Care: Women randomized to the control group will receive enhanced usual care (EUC). The World Health Organization (WHO) recommends 8 antenatal visits for a positive pregnancy experience, the number of visits our EUC control group participants will receive (depending on their gestational week). Usual care will also be enhanced by hospital staff receiving additional training in mental health treatment and counseling. Transportation will be facilitated to assist participants in attending appointments and medically indicated ultrasounds will be paid for (as in the intervention group).
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy (CBT) Intervention for Anxiety | Enhanced Usual Care
Started | 600 | 600
Completed | 380 | 375
Not Completed | 220 | 225

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy Intervention for Anxiety | Enhanced Usual Care | Total
Number analyzed (Participants) | 600 | 600 | 1200
Age, Continuous [Mean (Full Range); unit: Years] | 25.08 [18 to 40] | 25.46 [18 to 40] | 25.3 [18 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 600 | 600 | 1200
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 600 | 600 | 1200
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Pakistan | 600 | 600 | 1200
Baseline Hospital Anxiety and Depression Score (HADS) of >=8 on the anxiety subscale [Number; unit: participants] | 600 | 600 | 1200

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Combined Common Mental Disorders (CMDs, i.e. Anxiety and Depression).
Description: Data reported is the number of participants with Common Mental Disorders (CMDs), which is defined as a woman having either high anxiety or clinical depression at the time of follow-up. Both CMDs, anxiety was indicated by moderate to severe symptoms on the anxiety portion of the Hospital and Anxiety Scale (HADS). A cutoff of >10 was used as the threshold for moderate to severe levels of anxiety. A Major Depressive Episode (MDE) was measured with the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders (SCID), which is a semi-structured interview used to make major Axis I Diagnostic and Statistical Manual of Mental Disorders (DSM) diagnoses. Its scoring will be based on case or non-case basis.
Time Frame: 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Groups:
- Enhanced Usual Care: Women randomized to the control group will receive enhanced usual care (EUC). The World Health Organization (WHO) recommends 8 antenatal visits for a positive pregnancy experience, the number of visits our EUC control group participants will receive (depending on their gestational week). Reminders were given, provider visits facilitated (shorter wait times), and transportation to assist participants in attending appointments and medically indicated ultrasounds were paid for (as in the intervention group).
Arm/Group | Cognitive Behavioral Therapy Intervention for Anxiety | Enhanced Usual Care
Number analyzed (Participants) | 600 | 600
Participants | 57 | 178

2. Secondary Outcome: Number of Preterm Births
Description: Number of infants born with <37 weeks' gestation
Time Frame: at birth
Population: The analysis for the secondary outcomes on children is 720 rather than 755 for the primary outcome on mothers. The reason for this is because the sample size differed for these two groups for a number of reasons (e.g. women who did not carry their pregnancies to term).
Measure: Number; unit: infants
Arm/Group | Cognitive Behavioral Therapy Intervention for Anxiety | Enhanced Usual Care
Number analyzed (Participants) | 362 | 358
infants | 79 | 68

3. Secondary Outcome: Small-for-gestational Age Birth
Description: <10th% for gestational age at birth compared to the reference population
Time Frame: at birth
Population: as for outcome 2
Measure: Number; unit: infants
Arm/Group | Cognitive Behavioral Therapy Intervention for Anxiety | Enhanced Usual Care
Number analyzed (Participants) | 362 | 358
infants | 89 | 105

4. Secondary Outcome: Low Birthweight
Description: weight of ≤2500 grams
Time Frame: at birth
Population: as for outcome 2
Measure: Number; unit: infants
Arm/Group | Cognitive Behavioral Therapy Intervention for Anxiety | Enhanced Usual Care
Number analyzed (Participants) | 362 | 358
infants | 46 | 53

ADVERSE EVENTS:
Time Frame: 5 months
Description: None of the participants died, only there were some neo-natal deaths which were reported as Severe Adverse Event.
Arm/Group | Cognitive Behavioral Therapy Intervention for Anxiety | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/600 | 0/600
Serious Adverse Events (participants affected / at risk) | 48/600 | 42/600
Other Adverse Events (participants affected / at risk) | 0/600 | 0/600
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Therapy Intervention for Anxiety (N=600) | Enhanced Usual Care (N=600)
Serious Adverse Event (Injury, poisoning and procedural complications) | 48 (48) | 42 (42) — Still birth, miscarriage and child deaths

LIMITATIONS AND CAVEATS:
The Covid-19 pandemic occurred in the middle of data collection for this study. Because of the lockdowns data collection was halted for a period and also slowed. It probably also contributed to loss to follow up as many women were fearful of coming to the hospital.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT03880032/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT03880032/ICF_001.pdf